CLINICAL TRIAL: NCT05987280
Title: Development of a Core Outcome Set for Pharmacist-led Interventions in Chronic Kidney Disease: a Protocol for a Survey and e-Delphi Consensus Study
Brief Title: Core Outcome Set for Pharmacist-led Interventions in CKD
Acronym: COSP-KD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 40350
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Pharmacy; Pharmacist; Kidney disease; Core outcome set
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: We aim to use an online survey to collect data from participants. It is estimated that this survey will take 10 minutes to complete. The first part of the survey asks questions about the participant including what stakeholder group best describes them. The second part asks them about what outcomes are important in pharmacy research and in the management of kidney disease.
  Interventions: Other: eDelphi method
- Phase 2: The outcomes generated in this survey will be supplemented by outcomes identified in an ongoing systematic review being performed by our group. We will take this long list of outcomes and aim to reach consensus on a COS using a 2-round Delphi process. The Delphi process is a structured process used for forming a consensus, where stakeholder groups provide their opinions in an iterative approach for answering questions over several rounds.
  This will also take place using surveys online and we will submit an ethical amendment for each round with the questions and outcomes we will be seeking consensus on. In each Delphi round, participants will be asked to rate the importance of outcomes for inclusion or exclusion. Between each round, excluded outcomes will be removed. Included outcomes (those reaching consensus, defined as a minimum of 75% of participants who scored outcomes as agree or strongly agree or disagree or strongly disagree) will go into the COS.
  Interventions: Other: eDelphi method

INTERVENTIONS:
Other: eDelphi method — eDelphi method

SUMMARY:
Background Chronic kidney disease (CKD) is a progressive condition characterised by a gradual reduction in kidney function and structure over time. CKD is a risk factor for other morbidity, where it not only increases the likelihood of all-cause and cardiovascular mortality, but also can have a detrimental impact on quality of life. Whilst several systematic reviews have demonstrated the benefits of interventions delivered by pharmacists, there is significant variability in terms of the outcomes reported and an inconsistency with the measures used (e.g., medication adherence is often assessed using different outcome measures). The large heterogeneity of outcomes reported and the measures used in randomised controlled trials investigating the impact interventions involving pharmacists have on CKD patients makes it difficult to interpret findings and make comparisons between interventions have. This ultimately affects the quality of research and limits the ability to synthesize evidence, particularly in meta-analyses. Issues around inconsistent outcome reporting could be addressed with the development and application of agreed standardised sets of outcomes. Indeed, the significant range of outcomes in the CKD pharmacy literature led the authors in Raiisi et al., to state that further research is required to establish a core outcome set (COS) in CKD, in relation to pharmacy practice. COS are a collection of outcomes that are standardised and agreed upon, in which as a minimum, they should be measured and reported in all trials for a particular clinical topic. They are of importance as input is provided from a variety of stakeholders such as patients, researchers, family members, carers, and healthcare professionals, in which relevant outcomes are more likely to be identified, as well as helping reduce reporting bias and heterogeneity in the research literature. Currently no pharmacy-specific COS exists for interventions conducted in CKD.

Aims The overall objective is to develop a COS for clinical trials evaluating the efficacy or effectiveness of pharmacist-led interventions (i.e., interventions provided to patients are either pharmacist-led or involve their input) in people with CKD. The aim of Phase 1 is to conduct an online survey to explore outcomes of importance to stakeholders. The outcomes identified in Phase 1 will lead into a subsequent Delphi process to develop a COS (Phase 2).

Methods

Phase 1

The investigators aim to use an online survey to collect data from participants. The questions in this survey can be found in the attached documentation. It is estimated that this survey will take 10 minutes to complete. The first part of the survey asks questions about the participant including what stakeholder group best describes them. The second part asks them about what outcomes are important in pharmacy research and in the management of kidney disease.

Phase 2 The outcomes generated in this survey will be supplemented by outcomes identified in an ongoing systematic review performed by the research group. The investigators will take this long-list of outcomes and aim to reach a consensus on a COS using a 2-round Delphi process. The Delphi process is a structured process used for forming a consensus, where stakeholder groups provide their opinions in an iterative approach for answering questions over several rounds.

This will also take place using surveys online and the investigators will submit an ethical amendment for each round with the questions and outcomes we will be seeking consensus on. In each Delphi round, participants will be asked to rate the importance of outcomes for inclusion or exclusion. Between each round, excluded outcomes will be removed.

Included outcomes (those reaching consensus, defined as a minimum of 75% of participants who scored outcomes as agree or strongly agree or disagree or strongly disagree) will go into the COS.

Following the Delphi survey, the investigators will conduct a consensus day. A sample of participants will be invited to discuss the findings and reach a consensus on the final COS.

ELIGIBILITY:
Inclusion criteria:

The stakeholders that will be invited to participate in this survey include: 1) self-defined pharmacists involved in the care of kidney patients and non-renal pharmacists; 2) self-defined researchers involved in CKD and pharmacy research; 3) self-defined nurses and physicians involved in CKD management; 4) self-defined people living with kidney disease; and 5) their carers and/or family members.

It is likely that participants will not fit into distinct homogeneous groups; for example, researchers may also be registered pharmacists. Participants will answer questions relevant to their group. All participants over the age of 18 will be invited to take part in the survey

Exclusion criteria:

Any participants not self-defined as one of the above five groups.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The stakeholders that will be invited to participate in this survey include: 1) pharmacists involved in the care of kidney patients and non-renal pharmacists; 2) researchers involved in CKD and pharmacy research; 3) nurses and physicians involved in CKD management; 4) people living with kidney disease; and 5) their carers and/or family members.
  It is likely that participants will not fit into distinct homogeneous groups; for example, researchers may also be registered pharmacists. Participants will answer questions relevant to their group. All participants over the age of 18 will be invited to take part in the survey
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Generation of longlist of outcomes | 8 weeks
  The first part of the survey asks questions about the participant including what stakeholder group best describes them. The second part asks them about what outcomes are important in pharmacy research and in the management of kidney disease. Outcomes suggested by the participants will be entered into a 'longlist' of outcomes for Phase 2.
Delphi Round 1 | 4 weeks
  We will take this long list of outcomes and aim to reach consensus on a COS using a 2-round Delphi process. The Delphi process is a structured process used for forming a consensus, where stakeholder groups provide their opinions in an iterative approach for answering questions over several rounds.
  In Delphi round 1, participants will be asked to rate the importance of outcomes for inclusion or exclusion. Participants will score outcomes on a 7-point Likert scale.
Delphi Round 2 | 4 weeks
  Between Rounds 1 and 2, excluded outcomes will be removed. Included outcomes are defined as those reaching consensus, defined as a minimum of 75% of participants who scored outcomes as agree or strongly agree or disagree or strongly disagree
  In Delphi round 2, participants will be asked to rate the importance of remaining outcomes for inclusion or exclusion. Participants will score outcomes on a 7-point Likert scale.
  Final included outcomes (those reaching consensus, defined as a minimum of 75% of participants who scored outcomes as agree or strongly agree or disagree or strongly disagree) will go into the COS.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Wilkinson, Leicester, Leicestershire, United Kingdom